CLINICAL TRIAL: NCT00307424
Title: Comparison of Auto-Continuous Positive Airway Pressure Device(Auto-CPAP) With Conventional Fixed CPAP in Chinese Patients With Obstructive Sleep Apnea (OSA)
Brief Title: Comparison Between Auto CPAP and Fixed CPAP in Chinese Patients With OSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: CRE-2004.258-T
Record Dates: First submitted 2006-03-27; First posted 2006-03-28 (Estimated); Last update posted 2006-03-28 (Estimated); Status verified 2004-08

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

INTERVENTIONS:
Device: AutoCPAP
Device: FixCPAP

SUMMARY:
AutoCPAP would lead to better compliance than FixCPAP

DETAILED DESCRIPTION:
A prospective, randomized crossover cohort. Study subjects consisted of patients newly diagnosed with obstructive sleep apnea (OSA) confirmed with sleep study. All are CPAP naïve.

Randomization:

Arm 1: auto CPAP sleep study then auto CPAP for 2 months Arm 2: fixed CPAP titration then fixed CPAP for 2 months

Then switch over to the other arm

Trial end after 4 months, compliance and other parameters would be compared between two arms as described in the endpoint session.

ELIGIBILITY:
Inclusion Criteria:

* All subjects should be CPAP naïve.
* OSA confirmed with sleep study
* Presence of daytime symptoms with excessive daytime sleepiness
* Age between 18 to 65
* RDI greater than 30
* Agreed to participate in trial with informed consent signed

Exclusion Criteria:

* Patients not suitable to nasal CPAP because of facial abnormality leading to poor mask fitting.
* Patients with known COPD with type II failure
* Patients with known heart failure.
* Patients with predominant central sleep apnea.
* Patients need bilevel positive airway pressure ventilation.
* Patients refusing to participate the trial.
* Patients have difficulty to follow up regularly.
* patients with untreated or under treatment of hypothyroidism

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2004-08; Study Completion 2005-06

PRIMARY OUTCOMES:
To compare the compliance of auto-CPAP and fixed CPAP in terms of CPAP usage hours.
To compare the clinical efficacy of auto-CPAP and fixed CPAP in terms of pressure level to abolish OSA, Epworth sleepiness scale and quality of life questionnaire.
To compare patient acceptance of the different type of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: To K Wang, FHKCP, Principal Investigator — Prince of Wales Hosptial
Locations (2):
- China (2):
  - North District Hospital, Hong Kong
  - Prince of Wales Hospital, Hong Kong

REFERENCES:
- [Derived] To KW, Chan WC, Choo KL, Lam WK, Wong KK, Hui DS. A randomized cross-over study of auto-continuous positive airway pressure versus fixed-continuous positive airway pressure in patients with obstructive sleep apnoea. Respirology. 2008 Jan;13(1):79-86. doi: 10.1111/j.1440-1843.2007.01138.x. PMID 18197915